CLINICAL TRIAL: NCT02834221
Title: Ultrasound-guided or Anatomical Femoral Venipuncture for Pulmonary Vein Isolation for Atrial Fibrillation Treatment
Brief Title: Ultrasound-guided Femoral Vein Accessibility, Safety and Time for Atrial Fibrillation Treatment
Acronym: ULTRA-FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kenichiro Yamagata (Other Government)
Responsible Party: Sponsor-Investigator, Kenichiro Yamagata, MD, PhD, Institute for Clinical and Experimental Medicine
Organization: Institute for Clinical and Experimental Medicine (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ULTRA-FAST
Record Dates: First submitted 2016-06-29; First posted 2016-07-15 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Atrial Fibrillation; Peripheral Vascular Disease; Vascular Access Complications
Keywords: Femoral vein puncture
MeSH Terms: conditions — Atrial Fibrillation; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real-time ultrasound-guided puncture (Experimental): Cannulate each femoral veins with two wires with real-time ultrasound-guided method.
  Interventions: Device: Real-time ultrasound-guided puncture
- Anatomical landmark guided puncture (Other): Cannulate each femoral veins with two wires with the anatomical landmark guided method.
  Interventions: Other: Anatomical landmark guided puncture

INTERVENTIONS:
Device: Real-time ultrasound-guided puncture — A 7 megahertz ultrasound linear probe will be used.
  Arms: Real-time ultrasound-guided puncture
Other: Anatomical landmark guided puncture — Anatomical landmark puncture
  Arms: Anatomical landmark guided puncture

SUMMARY:
This study is designed to evaluate the use of real-time ultrasound-guided femoral venipuncture during pulmonary vein isolation for treating atrial fibrillation .

DETAILED DESCRIPTION:
The number of pulmonary vein isolation (PVI) therapy for atrial fibrillation (AF) is increasing. Multiple femoral vein cannulation is mandatory for this procedure. There are mainly two methods to cannulate the femoral vein; by anatomical landmark or by under real-time ultrasound-guided. As high anticoagulant level is required for the procedure, there are 0-13% of vascular access complication.

Real-time ultrasound assistance for central venous catheter cannulation has been proven to reduce complications. In the field of AF treatment, multiple femoral vein cannulation is required as many catheter is required for the procedure and larger sheaths are inserted with a high anticoagulant level during the procedure. In this setting, the use of ultrasound use is not well studied.

The current study is to confirm whether real time ultrasound-guided femoral vein cannulation for PVI can prevent complications, reduce puncture time, puncture attempts and accidental artery puncture compared to conventional anatomical approach. Two seethes for each femoral vein is going to be cannulated.

The study design is a multicenter prospective randomized trial to compare the above safety and efficacy by using the ultrasound-guided and anatomical landmark approach. Also time for cannulation, number of puncture attempts, need of X-ray for cannulation will be analyzed in the setting of patient factors including age, body mass index and sex.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pulmonary vein isolation with radiofrequency catheter ablation for atrial fibrillation treatment.

Exclusion Criteria:

* Patients with prior known vascular access problems or priory included to the current study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2016-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Major complications | After the puncture up to 12 weeks
  Total patient number of vascular complications requiring surgical treatment, retroperitoneal hematoma requiring blood transfusion or hemoglobin drop of 3 >g/dl, strong pain at the groin, prolonging hospital stay and requiring hospital admission after discharge.

SECONDARY OUTCOMES:
Unsuccessful femoral vein cannulation | Immediately after the puncture
  Number of patients with unsuccessful femoral vein cannulation defined as crossing over to the other randomized method or change of operator to cannulate all wires.
Number of puncture attempts | Immediately after the puncture
  Number of puncture attempts to cannulate all wires.
Total puncture time | Immediately after the puncture
  Time from giving anesthesia to the groin till confirming all wires in the infra vena cava with the X-ray.
Number of artery mis-punctures | Immediately after the puncture
  Number of artery mis-punctures attempts to cannulate all wires.
Use of X-ray for successful wire cannulation | Immediately after the puncture
  If there is a need of X-ray to cannulate the wire into the infra vena cava.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Kautzner, MD, PhD, Study Director — Institute for Clinical and Experimental Medicine
Locations (4):
- Czechia (3):
  - Regional Hospital Liberec, Liberec
  - Institute for Clinical and Experimental Medicine, Prague
  - Ústřední vojenská nemocnice, Prague
- Kawakita General Hospital, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yamagata K, Wichterle D, Roubicek T, Jarkovsky P, Sato Y, Kogure T, Peichl P, Konecny P, Jansova H, Kucera P, Aldhoon B, Cihak R, Sugimura Y, Kautzner J. Ultrasound-guided versus conventional femoral venipuncture for catheter ablation of atrial fibrillation: a multicentre randomized efficacy and safety trial (ULTRA-FAST trial). Europace. 2018 Jul 1;20(7):1107-1114. doi: 10.1093/europace/eux175. PMID 28575490